CLINICAL TRIAL: NCT03007901
Title: Mindful Climate Action: Improving Health While Reducing Carbon Footprint: A Pilot Study
Brief Title: Mindful Climate Action: Improving Health While Reducing Carbon Footprint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-1336
Record Dates: First submitted 2016-12-13; First posted 2017-01-02 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilot Cohort 1 (Experimental): This Pilot Study will be conducted to allow us to evaluate and test the various study processes, including: consent/enrollment, run-in-trial monitoring, measurement tools, outcome assessment, educational materials, and especially the mindfulness-based climate action trainings. The pilot study does not include a control group, and data will not be used for efficacy outcome analysis.
  Interventions: Behavioral: Mindful Climate Action

INTERVENTIONS:
Behavioral: Mindful Climate Action — Educational and Behavioral Training Curriculum: An article describing our proposed program was recently published in Sustainability (1) and is summarized here. Experienced instructors from the UW Integrative Medicine Mindfulness Program will teach the 8-week program. Classes will meet weekly for 2½ hours, with a 6 hour weekend retreat. Twenty to 45 minutes of daily home practice will be guided by audio recordings leading participants through body scan, sitting meditations, breath awareness, and mindful movement. Each of the 2½ hour weekly classes includes topics (~30 min) relating to climate change, energy use, and carbon footprint.
  Other Names: MBSR with Climate Education

SUMMARY:
To work with community partners to pilot test a mindfulness-based behavioral program aimed at: (a) enhancement of health and well-being, and (b) reduction in carbon footprint; (2) to develop, implement, and refine methods for assessing carbon footprint at the individual level; and (3) to work with pilot participants and community partners to carry out a proof-of-concept research study to assess impact on health, well-being, and carbon footprint.

DETAILED DESCRIPTION:
This Pilot Study will be conducted to allow us to evaluate and test the various study processes, including: consent/enrollment, run-in-trial monitoring, measurement tools, outcome assessment, educational materials, and especially the mindfulness-based climate action trainings. The pilot study does not include a control group, and data will not be used for efficacy outcome analysis. The investigators anticipate doing two pilot cohorts of roughly 16 persons/group. The pilot cohorts will not be simultaneous.

Participants will meet for 2½ hour sessions, once per week for eight weeks. An additional 6-hour retreat will be scheduled over a weekend towards the end of the program. Participants will receive about 26 hours of contact time. Their daily home practice will be guided by audio recordings (25 to 45 minutes) that lead them through their formal meditation practice of the body scan, sitting meditations, and gentle yoga. Participants will be asked to practice for 5 or 6 days per week at home, using these audio recordings or on their own. They will also be asked to select a daily practice time that works best for them, perhaps early morning, after work, or later in the evening. Participants will record what they practice and for how long either on paper log sheets or using a web-based data form.

Climate change, energy, and carbon footprint knowledge will be assessed by a college intro-level test (pre- and post-training). Electrical and gas use will be assessed directly by inspecting Madison Gas and Electric (MG&E) utility records. Miles driven in automobile will be assessed by self-report, verified with odometer readings of primary vehicle done by study staff. Active transportation and motor vehicle travel will be measured using a free, smart phone app called MOVES. In order to extract the activity data from the user's phone, each participant will download another free app called TRAQS CSV Exporter (https://labs.traqs.me/moves/) which will export data once monthly over the course of the year. Individual movement/transportation activity data obtained from this app will provide the study team with data allowing an in-depth and fine-grained understanding of transportation behaviors across the study time period.

Dietary composition will be assessed by validated dietary recall, with proportion of dietary calories from animal versus plant sources as the primary assessment. Composite carbon footprints will be calculated. In addition to carbon footprint, the investigators will be assessing health co-benefits, including several domains of mental and physical health (validated self-report measures) and active transport assessed using Actigraph accelerometers.

Participants will be asked to provide feedback through interviews regarding the curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 65 years at enrollment will be assessed by self-report and date of birth. This relatively broad age range will facilitate enrollment and will enhance generalizability of results. This range will also tend to include people with moderate to large carbon footprints, possibly allowing room for measurable improvement with mindfulness training.
* Fluency in English (oral, reading, and writing) is necessary to complete all study parameters including: providing consent, completion of questionnaires and online surveys, and intervention objectives.
* Willingness and ability to carry out all study-specific tasks, including commitment to provide data, wear an ActiGraph for one week twice over the course of the study, and be monitored throughout the research study period.
* Participants must be owners (or co-owners) of single family dwelling, and must have been in the same location for the prior 12 months, with no expectation of moving during the study. Utility service to the single family dwelling must be provided by MG&E (gas and electric) and Madison Water Utility. This is necessary to accurately assess and compare household energy and water use across participants and randomized groups.
* Participants must own (or co-own or lease) an automobile and drive it at least 5000 miles per year (assessed by self-report). The choice of 5,000 miles as cutoff is arbitrary, but will exclude those who do not drive much, and would therefore have less capacity for measureable improvement. People who share the use of a car with no more than one other person but who drive the majority of miles will be included, as will people who own and drive two primary vehicles. People who own and regularly drive more than two vehicles will be excluded due to the added participant and staff burden involved with obtaining odometer readings.
* Ownership, use, and familiarity with a smart phone (either iPhone or Android type) will be required due to planned use of the MOVES app to obtain major outcome data.
* Only one member per household will be allowed to participate.

Exclusion Criteria:

* Participants will be excluded if they currently or recently participate in meditative practice or mindfulness or other meditation training in the past 3 years. Assessed by answering "Yes" to any of the following questions: Do you meditate on a regular basis? In the last year, have you meditated at least weekly for 2 or more months in a row? Have you received meditation training in the last 5 years? Have you taken part in a mindfulness class or mindfulness sessions during the past 5 years?
* People with self-described vegan or vegetarian diets (self-assessed average meat ingestion frequency less than once/week) will be excluded, as one goal of the trainings is to influence dietary habits away from meats (especially beef) and towards vegetables and other plant-based foods. Only those who answer "Yes" to "Do you tend to eat at least one meal with some meat in it on most days of the week?" will be eligible to participate.
* People with serious physical, medical, or mental condition precluding adherence to study protocol will be excluded. Questionable cases will be reviewed by the study physicians.
* Those that are unable/unwilling to successfully complete baseline assessment, including in-person meetings, data-collection, and other tasks will be excluded from the study. Inability to complete a sample of the study requirements will indicate an inability to complete full study requirements.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01; Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Estimated carbon footprint | 6 months
  Carbon footprint (CF) will be estimated. Individual-level carbon footprints (ICF) are assessed as ICF = ΣCiEi where each term is the product of the degree of consumption (C) and the CO2 equivalent radiative forcing emission (E) of that input (i). Greenhouse gas emission (E) weightings applied to individual consumption levels (C) will be expressed in metric tons CO2-equivalent/year (CO2e).

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Barrett, MD PhD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett B, Grabow M, Middlecamp C, Mooney M, Checovich MM, Converse AK, Gillespie B, Yates J. Mindful Climate Action: Health and Environmental Co-Benefits from Mindfulness-Based Behavioral Training. Sustainability. 2016 Oct;8(10):1040. doi: 10.3390/su8101040. Epub 2016 Oct 17. PMID 28008371